CLINICAL TRIAL: NCT04110067
Title: Clinical Results of Small Incision Lenticule Extraction (SMILE) for the Correction of High Myopia
Status: Recruiting | Type: Observational
Sponsor: Suphi Taneri (Other)
Responsible Party: Sponsor-Investigator, Suphi Taneri, Director, St. Franziskus Hospital
Organization: St. Franziskus Hospital (Other)
Other Study IDs: SMILE > 7.75D
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Myopia; High Myopia
Keywords: Myopia; Refractive Surgery; Small Incision Lenticule Extraction; SMILE
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- 1: SMILE - Correction of eyes with myopia of more than -7.75 D
  Interventions: Other: Small Incision Lenticule Extraction (SMILE) with Visumax (Carl Zeiss Meditec, Jena)

INTERVENTIONS:
Other: Small Incision Lenticule Extraction (SMILE) with Visumax (Carl Zeiss Meditec, Jena) — Creation of a corneal tissue disk called lenticule and extraction through a minimally invasive incision, utilizing only a femtosecond laser
  Other Names: RelaxSmile

SUMMARY:
Small Incision Lenticule Extraction (SMILE) was introduced in 2011 using the VISUMAX femtosecond laser (Carl Zeiss Meditec, Jena, Germany). It is designed for correction of myopia and myopic astigmatism.

It involves the creation of a corneal tissue disk called lenticule and its extraction through a minimally invasive incision, utilizing only a femtosecond laser. This enables rapid visual recovery with very little discomfort to the patient.

This observational case series monitors visual and refractive outcomes of myopic correction for more than -7.75 D.

It is to

* gather long-term results and refractive stability
* detect rare complications or side-effects
* evaluate the efficacy in a large number of patients

ELIGIBILITY:
Inclusion Criteria:

* adults
* myopia more than -7.75 D
* refractive stability more than 1 year

Exclusion Criteria:

* corneal irregular astigmatism
* ectatic conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with myopia more than -7.75 D seeking refractive surgery
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Subjective Distance Refraction | 1 year
  Subjective Refraction
Distance Visual Acuity | 1 year
  Visual Acuity sine and cum correctione

SECONDARY OUTCOMES:
Tectonic stability as assessed by Pentacam | 1 year
  Corneal tectonic stability post surgery as assesed by Scheimpflug-Tomography
Epithelial thickness map in Optical coherence tomography | 1 year
  Change of Thickness of epithelium pre and post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Suphi Taneri, MD, Study Chair — Center for Refractive Surgery Muenster
Locations (1):
- Center for Refractive Surgery, Münster, North Rhine-Westphalia, Germany